CLINICAL TRIAL: NCT05326594
Title: Effects of Physical Therapy on Improving Disc Height Index, Postural Stability, Pain and Function in Persons With Discogenic Low Back Pain
Brief Title: Effects of Physical Therapy on Improving Disc Height, Postural Stability, Pain and Function in Persons With Discogenic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/5
Record Dates: First submitted 2022-03-29; First posted 2022-04-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain; Disk Prolapse
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Therapy (Experimental)
  Interventions: Procedure: Mckenzie Extension Protocol; Procedure: Lumbar SNAGs; Device: Inferential therapy; Procedure: Heat Therapy

INTERVENTIONS:
Procedure: Mckenzie Extension Protocol — Mckenzie Extension Exercise Protocol will be performed by participants in prone position
Procedure: Lumbar SNAGs — Lumbar SNAGs will be performed in lumbar flexion and extension in standing Position
Device: Inferential therapy — 4 pole inferential therapy in combination with superficial heating for 20 minutes
Procedure: Heat Therapy — superficial heating for 20 minutes

SUMMARY:
Lumbar degenerative disc disease and discogenic low back pain is comparatively common and disabling musculoskeletal condition, however there is no conclusive evidence regarding the positive effects of conservative physical therapy management in terms of radiological changes and improvement in disc height. For this reason, the current study will not only look into the positive effects of conservative physical therapy on postural stability, pain and function, but also in terms of disc height in persons with discogenic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants
* Aged 18-50 years old
* low back pain intensity less than 80/100mm on visual analogue scale
* positive centralization phenomenon
* low signal intensity of IV disc on T2 - weighted MRI
* high intensity zone towards the posterior aspect of the disc on MRI

Exclusion Criteria:

* Individuals with and any musculoskeletal, metabolic, or neurological disorders that may impair gait, postural stability or sensory integrity will be excluded from the study.

Ages: 18 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Back Pain | 2 weeks
  Pain will be measured via Visual Analogue Scale. A higher score signifies poor outcome.
Lumbar Range of Motion | 2 weeks
  Lumbar Range of Motion will be measured via inclinometer. A higher score signifies good outcome.
Postural Stability | 2 weeks
  Postural Stability will be measured via Biodex Balance System. A higher score signifies poor outcome.
Lumbar Disability | 2 weeks
  Disability will be measured via Oswestry Disability Index.
Step length | 2 weeks
  Step length during gait will be analyzed using observational gait analysis. A greater step length signifies better outcome
Stride length | 2 weeks
  Stride length during gait will be analyzed using observational gait analysis. A greater stride length signifies better outcome
Gait velocity | 2 weeks
  Velocity during gait will be analyzed using observational gait analysis. A greater gait velocity signifies better outcome
Disc Height | 2 weeks
  Disc will be analyzed using Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Osama, PhD*, Principal Investigator — FUI; Aamer Naeem, PhD*, Principal Investigator — FUI
Locations (1):
- Foundation University Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osama M, Naeem A, Tariq S, Mushtaq S, Siddiqi FA, Afridi S. Effects of physical therapy on improving disc height index, postural stability, pain and function in persons with discogenic low back pain. J Pak Med Assoc. 2025 Mar;75(3):378-382. doi: 10.47391/JPMA.20384. PMID 40143467